CLINICAL TRIAL: NCT06188845
Title: Improved Hand Function in High-functioning Stroke Survivors by Applying Kinesio Taping: A Prospective Clinical Trial
Brief Title: Kinesio Taping in Stroke Patient
Acronym: Kinesio taping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taiwan Municipal An-Nan Hospital-China Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TMANH108-REC009; TMANH108-REC009 (Other: institutional review board of Taiwan Municipal An Nan Hospital-China Medical University)
Record Dates: First submitted 2023-09-12; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Stroke; Cardiovascular Diseases; Physical Disability
Keywords: kinesio tape; high-functioning stroke; hand function; stroke
MeSH Terms: conditions — Stroke; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KT group (Experimental): Participants in the KT group were applied I-shaped Kinesio tape to the wrist extensor and pronator teres of the hemiplegic forearm for 2 days. Throughout the 2-day experiment, all participants received regular conventional rehabilitation.
  Interventions: Other: Kinesio taping
- CT group (No Intervention): Participants in the CT group did not receive tape intervention but received regular conventional therapy.

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping is a non-invasive physical treatment, which is breathable, hypoallergenic and elastic. Because of the mechanical properties and physiological effects, Kinesio taping has been thought to relieve pain, reduce swelling, support and relax soft tissue, promote motor performance, and correct posture or abnormal movement patterns.
  Arms: KT group

SUMMARY:
Despite being nearly independent in daily life, chronic high-functioning stroke survivors still experienced mild impairments in skilled hand function. Kinesio Taping (KT) has been used to help stroke patients improve their balance and ambulation. Few studies explored the effects of KT on fine motor function in stroke patients. The purpose of this study was to investigate the hand function performance of high-functioning stroke survivors after KT. Participants were divided into two groups: KT group and control group. Last two days, the KT group received KT intervention. After the taping was removed, baseline and post-test evaluation were conducted. Outcome measures included muscle strength, range of motion (ROM), spasticity, fine motor function, and self-reported upper limb disability. The results revealed that the KT group had less spasticity, increasing ROM trend, and improved fine motor function and disability. KT improved spasticity, active movement, and muscle flexibility, resulting in more skilled and delicate hand function in chronic high-functioning stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

* (1) Stroke with unilateral hemiparesis, (2) onset duration > 6 months, (3) Brunnstrom stage in the proximal and distal parts of the upper extremity > stage III, and (4) adequate cognitive ability to understand and cooperate with the experiment procedure.

Exclusion Criteria:

* Participants with skin problem (such as allergies, open wound), a history of upper extremity musculoskeletal diseases (such as fractures, tendon ruptures), or other peripheral neurological or systemic diseases were excluded.

Ages: 32 Years to 77 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2021-01-04 (Actual); Primary Completion 2022-02-09 (Actual); Study Completion 2022-02-09 (Actual)

PRIMARY OUTCOMES:
Muscle strength | Baseline and post-test( 2 days later)
  The maximum grip force and the muscle strength of the wrist extensor and flexor
AROM and PROM | Baseline and post-test( 2 days later)
  The AROM and PROM of wrist flexion and extension (AROM and PROM in degrees). The AROM and PROM of the wrist flexion and extension were measured with the goniometers.
Spasticity | Baseline and post-test( 2 days later)
  Spasticity of wrist and finger flexor and extensor. The spasticity of wrist and finger flexor and extensor were assessed with modified Ashworth Scale (MAS).
The Action Research Arm Test | Baseline and post-test( 2 days later)
  gross motor and fine motor function of the upper limb, which included grasp, grip, pinch, and gross movement
Quick DASH | Baseline and post-test( 2 days later))
  To measure the disability and symptoms of the upper limb, participants self-reported the Disability of the Arm, Shoulder and Hand (Quick DASH) questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ya-Wen Tsai, MS, Principal Investigator — Department of Rehabilitation, An Nan Hospital, China Medical University, Tainan, Taiwan
Locations (1):
- An Nan Hospital, China Medical University, Tainan, Taiwan